CLINICAL TRIAL: NCT05569473
Title: Clinical and Radiographic Evaluation of Volume Stable Collagen Matrix (VCMX) in the Regenerative Outcome of Periodontal Intrabony Defects in Humans: a Randomized Controlled Clinical Trial."
Brief Title: Evaluation of Volume Stable Collagen Matrix in the Regenerative Outcome of Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pratiksha PGIDS/BHRC/22/30
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Intrabony defect filled with VCMX after along with open flap debridement [OFD+VCMX])
  Interventions: Procedure: TEST GROUP: VCMX + OFD, CONTROL GROUP : OFD ONLY
- control group (Experimental): OFD will be done and After this, flaps would be approximated and sutured at the original position with a monofilament suture material using interrupted sutures.
  Interventions: Procedure: TEST GROUP: VCMX + OFD, CONTROL GROUP : OFD ONLY

INTERVENTIONS:
Procedure: TEST GROUP: VCMX + OFD, CONTROL GROUP : OFD ONLY — A full-thickness mucoperiosteal flap will be raised, no bone recontouring would be performed, Thorough debridement of the surgical site would be performed. For the test group, VCMX would be placed according to the dimensions of the intrabony defect after open flap debridement (OFD). For the control group, OFD will be done and After this, flaps would be approximated and sutured at the original position with a monofilament suture material using interrupted sutures.

SUMMARY:
Periodontal intrabony defect is a specific osseous defect with definite morphology. Numerous therapeutic modalities for restoring such defects have been investigated.

Nanocomposites and nanostructured materials are thought to have a key function in hard tissue research, since natural bone tissue is a distinctive model of a nanocomposite. Collagen has been potentially used in periodontal tissue engineering. The integration of collagen as a structural protein, serving as an essential component of connective tissue into three-dimensional scaffolds implanted after periodontal injury, necrosis or inflammation has attracted much attention in tissue regeneration. If a collagen matrix collapses after implantation, host cell migration and blood vessel penetration may be impaired, which in turn negatively influences tissue degradation and integration as well as extracellular matrix production in the interior of the biomaterial. Thus, volume stability is an important parameter for tissue augmentation.

Volume stable collagen matrix (VCMX) is able to overcome the volume stability limitation of most commercially available grafts.7 It is one of the most biocompatible, novel material to be used in this study. It will be the first time that VCMX is to be used to regenerate the periodontal tissues in intrabony defects in humans.

DETAILED DESCRIPTION:
Periodontal intrabony defect is a specific osseous defect with definite morphology. Numerous therapeutic modalities for restoring such defects have been investigated.

Nanocomposites and nanostructured materials are thought to have a key function in hard tissue research, since natural bone tissue is a distinctive model of a nanocomposite. Collagen has been potentially used in periodontal tissue engineering. The integration of collagen as a structural protein, serving as an essential component of connective tissue into three-dimensional scaffolds implanted after periodontal injury, necrosis or inflammation has attracted much attention in tissue regeneration. If a collagen matrix collapses after implantation, host cell migration and blood vessel penetration may be impaired, which in turn negatively influences tissue degradation and integration as well as extracellular matrix production in the interior of the biomaterial. Thus, volume stability is an important parameter for tissue augmentation.

Volume stable collagen matrix (VCMX) is able to overcome the volume stability limitation of most commercially available grafts. It is one of the most biocompatible, novel material to be used in this study. While mechanical stability is achieved by chemical crosslinking, mechanical testing demonstrated preserved elasticity of the material over 14 days. It has shown quite impressive results in resolving the intrabony defects in animal studies with an average of 58.56% of new bone formation . Sustained release of growth factors with preserved biological activity is one of its important properties. It will be the first time that VCMX is to be used to regenerate the periodontal tissues in intrabony defects in humans.

MATERIAL AND METHODS:

Systemically healthy forty chronic periodontitis (stage II and III periodontitis) patients having 40 intrabony defects will be randomly assigned into test group (intrabony defect filled with VCMX after open flap debridement [OFD+VCMX]) and control group (OFD only). Patients fulfilling the eligibility criteria will be enrolled in the trial after obtaining informed consent. Primary outcome measures include probing pocket depth, clinical attachment level, and percentage bone fill (%BF). All parameters will be recorded at baseline,3,6 and 9 months postsurgical follow-up.

This study will be conducted at Department of Periodontics and Oral Implantology, PGIDS, Rohtak, Haryana. It is a Randomized controlled clinical trial which is to be carried out with a follow up period of 9 months. It has been approved by the institutional review board and institutional ethical committee.

Parameters recorded for experimental and adjacent teeth will include: PIaque index (PI) and Gingival Index (GI), bleeding on probing (BOP, %), PPD, CAL, and gingival recession (REC). Parameters that will be assessed using CBCT will include defect fill (DF), alveolar crest changes (ACC), and defect resolution (DR). Each patient will receive the initial phase of the therapy, which will include oral hygiene instructions, supragingival and subgingival debridement. Periodontal re-evaluation will be done to confirm the sites that required surgical therapy. A full-thickness mucoperiosteal flap will be raised, no bone recontouring would be performed, Thorough debridement of the surgical site would be performed. For the test group, VCMX would be placed according to the dimensions of the intrabony defect after open flap debridement (OFD). For the control group, OFD will be done and After this, flaps would be approximated and sutured at the original position with a monofilament suture material using interrupted sutures. Periodontal dressing (Coe-Pak, GC) will be used to cover and protect the surgical area. All study participants will be prescribed amoxycillin 500 mg (Mankind Pharmaceuticals) three times daily for 5 days and ibuprofen 400 mg (Abbott India) three times daily for 3 days. Patients will be instructed to rinse twice daily with 0.12% chlorhexidine. Patients will not be advised to use mechanical means of plaque control in the surgical area until sutures were removed. Sutures and periodontal dressing will be removed after a 1-week postoperative interval. Instructions for maintenance of proper oral hygiene will be reinforced.

ELIGIBILITY:
Inclusion Criteria:

Two-, three-, or combined two/three-wall intrabony defects with depth ≥ 3 mm (initially analyzed by transgingival probing and intraoral periapical radiographs and confirmed after flap elevation)

* PPD ≥ 5 mm
* CAL ≥ 3 mm
* tooth mobility < grade 1
* experimental teeth and adjacent teeth would be required to be vital and free of caries or dental restorations.

Exclusion Criteria:

* Any systemic illness that could affect the periodontium or outcome of periodontal therapy
* patients on medications such as corticosteroids or calcium channel blockers
* long-term nonsteroidal anti-inflammatory drug therapy
* pregnant or lactating women
* current and past smoker
* Periodontitis stage 4
* teeth with one-wall defect, the presence of exostoses and ledges, grade II and grade III mobile teeth, defects extending to a root furcation area, unrestorable teeth, fractured/perforated roots, developing permanent teeth, endodontically treated teeth, and teeth with premature contact and dental prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) | 9 MONTHS
  probing depth will be measured as the distance from the gingival margin to the base of pocket the probing depth. Measurements will be assessed using a calibrated manual periodontal probe (PCP UNC-15 Hu friedy Chicago, IL, USA. The probe will be inserted in the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of a tooth mesio buccal, mid buccal, distobuccal, mesio lingual, mid lingual and distolingual measurements will be rounded to the nearest whole mm.
Clinical attachment level (CAL) | 9 MONTHS
  clinical attachment level will be measured at the distance between the base of the pocket and the cement enamel junction (CEJ). Measurements will be made at 6 sites of each tooth - mesiobuccal, mid buccal, disto buccal, mesio lingual, mid lingual and distolingual using UNC 15 probe.
BONE FILL PERCENTAGE(BF%) | 9 MONTHS
  bone fill percentage will be recorded pre op and post op.

CONTACTS AND LOCATIONS:
Overall Officials: Pratiksha Chordiya, MDS, Principal Investigator — Postgraduate Institute of Dental Sciences Rohtak
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No